CLINICAL TRIAL: NCT01134484
Title: A Phase 3, Prospective, Randomized Clinical Study of VELCADE-Thalidomide-Dexamethasone (VTD) Versus Thalidomide-Dexamethasone (TD) for Previously Untreated Multiple Myeloma (MM) Patients Who Are Candidates to Receive Double Autologous Transplantation
Brief Title: VELCADE-Thalidomide-Dexamethasone (VTD) vs Thalidomide-Dexamethasone (TD) Incorporated Into Double Autotransplantation for Untreated Multiple Myeloma (MM)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michele Cavo (Other)
Collaborators: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor-Investigator, Michele Cavo, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-BO2005; 2005-003723-39 (EudraCT Number); 26866138-MMY-3006 (Other Grant/Funding Number: Janssen-Cilag SpA)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Multiple Myeloma
Keywords: autologous stem cell transplantation; complete remission; bortezomib; thalidomide; progression free survival; induction and consolidation therapy
MeSH Terms: conditions — Multiple Myeloma; Pathologic Complete Response | interventions — Bortezomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VTD (Experimental)
  Interventions: Drug: Velcade; Drug: Thalidomide; Drug: Dexamethasone; Procedure: Peripheral Blood Stem Cell (PBSC) collection; Procedure: First Autologous Transplantation; Procedure: Second Autologous Transplantation
- TD (Active Comparator)
  Interventions: Drug: Thalidomide; Drug: Dexamethasone; Procedure: Peripheral Blood Stem Cell (PBSC) collection; Procedure: First Autologous Transplantation; Procedure: Second Autologous Transplantation

INTERVENTIONS:
Drug: Velcade — * INDUCTION THERAPY: 1.3 mg/sqm as a bolus i.v. injection on days 1, 4, 8 and 11 (3 courses, 21 days each)
  * REMISSION CONSOLIDATION THERAPY: 1.3 mg/sqm as a bolus i.v. injection on days 1, 8, 15 and 22 (2 courses, 35 days each)
  Other Names: Bortezomib
  Arms: VTD
Drug: Thalidomide — * INDUCTION THERAPY: 100 mg/d on days 1-14, 200 mg/d on days 15-63 (in case of delay of HD-CTX , Thalidomide will be continued until the day before Cyclophosphamide as priming therapy for PBSC collection)
  * AFTER PBSC COLLECTION: 100 mg/d from day after last PBSC collection until the day before first course of MEL-200
  * AFTER FIRST TRANSPLANTATION: 100 mg/d from recovery of hematopoiesis until the day before the second course of MEL-200
  * REMISSION CONSOLIDATION THERAPY (starting 3 months after the second autologous transplantation): 100 mg/d days 1-70
  Other Names: Talidomide
Drug: Dexamethasone — * INDUCTION THERAPY
    1. VTD ARM: 40 mg/d days 1-2, 4-5, 8-9 and 11-12 (3 cycles, 21 days each)
    2. TD ARM: 40 mg/d days 1-4 and 9-12 (3 cycles, 21 days each)
  * AFTER PBSC COLLECTION: 40 mg/d for 4 days (starting the same day of resumption of Thalidomide)
  * AFTER FIRST TRANSPLANTATION: 40 mg/d for 4 days (starting the same day of resumption of Thalidomide) and repeated every 28 days, for 3 months
  * REMISSION CONSOLIDATION THERAPY (starting 3 months after the second autologous transplantation)
    1. VTD ARM: 40 mg/d days 1-2, 8-9, 15-16 and 22-23 (2 cycles, 35 days each)
    2. TD ARM: 40 mg/d days 14 and 20-23 (2 cycles, 35 days each)
  Other Names: Soldesam
Procedure: Peripheral Blood Stem Cell (PBSC) collection — * Cyclophosphamide (CTX): 4 g/sqm given in a single day (day 0)
  * G-CSF: 10 µcg/kg/d, starting on day +2 from CTX and continuing until completion of PBSC collection
Procedure: First Autologous Transplantation — * HIGH-DOSE MELPHALAN (MEL-200): 200 mg/sqm, given as a single dose i.v. (day -2) followed by PBSC infusion 48 hours later (day 0)
  * G-CSF: 5 µcg/kg daily starting from day +6 after grafting and continuing until the patient's ANC is more than 0.5x10^9/L for 3 consecutive days
Procedure: Second Autologous Transplantation — * HIGH-DOSE MELPHALAN (MEL-200): 200 mg/sqm, given as a single dose i.v. (day -2) followed by PBSC infusion 48 hours later (day 0)
  * G-CSF: 5 µcg/kg daily starting from day +6 after grafting and continuing until the patient's ANC is more than 0.5x10^9/L for 3 consecutive days

SUMMARY:
Thalidomide-Dexamethasone (TD) is a standard induction therapy for Multiple Myeloma (MM). The present study is designed to compare TD with VELCADE-Thalidomide-Dexamethasone (VTD) as induction therapy in preparation for, and as consolidation after, melphalan-based double autologous stem cell transplantation for previously untreated patients aged ≤65 years with symptomatic MM. Primary study endpoint is the rate of complete response (CR) plus near-complete response (nCR) to induction treatment. Secondary endpoints include the rate of CR plus nCR to double transplantation and subsequent consolidation therapy, time to progression (TTP), progression-free survival (PFS),overall survival (OS) and toxicity profile of both VTD and TD.

DETAILED DESCRIPTION:
This prospective phase 3 trial is aimed at evaluating whether, in comparison with standard TD, addition of Velcade to TD increases rate of CR and nCR from 15% to 30%, respectively. For this purpose, symptomatic patients aged 18-65 years with previously untreated MM and quantifiable M-protein in serum or urine are randomized (1:1) to receive induction therapy comprising three 3-week cycles of Velcade 1.3 mg/sqm, days 1, 4, 8, 11, thalidomide 100 mg, days 1-14, cycle 1, then 200 mg daily, and dexamethasone 40 mg, days 1, 2, 4, 5, 8, 9, 11, 12, or thalidomide and dexamethasone (same schedule and dosage as in VTD). Randomization to VTD or TD is stratified according to International Staging System disease stage at diagnosis. Following induction therapy, patients in both arms receive cyclophosphamide (4 g/sqm, day 0 and granulocyte colony-stimulating factor, 10 μcg/kg/day, from day +2) to collect autologous peripheral blood stem cells (minimum threshold CD34+ cells: 4 x 10^6/kg) and two subsequent courses of stem cell-supported high dose melphalan (200 mg/sqm), 3 to 6 months apart. Upon neutrophil (≥1 x 10^9/L) and platelet (≥75 x 10^9/L) recovery following the first autotransplantation, patients receive thalidomide (100 mg daily) and dexamethasone (40 mg, days 1-4 every 4 weeks) as bridge therapy until the day before the second transplantation.

Patients initially randomized to receive VTD or TD induction therapy are planned to receive two 5-week cycles of VTD (Velcade 1.3 mg/sqm, days 1, 8, 15, 22; thalidomide 100 mg daily; dexamethasone 40 mg, days 1, 2, 8, 9, 15, 16, 22, 23) or TD (thalidomide 100 mg daily; dexamethasone 40 mg, days 1-4 and 20-23) as consolidation therapy, starting 3 months after last transplant. Maintenance therapy comprise dexamethasone 40 mg, days 1-4, repeated monthly until relapse or progression.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of symptomatic MM based on standard criteria.
* No prior or current systemic therapy for MM, including steroids.
* At least 18 years and less than 65 years of age.
* Presence of quantifiable M protein in serum (e.g. greater than 1 g/dL for IgG MM, greater than 0.5 g/dL of IgA or IgD MM) or urine (e.g. greater than 200 mg/day for BJ MM).
* Karnofsky performance status (PS) at least 60%.
* Willing and able to comply with the protocol requirements.
* Agreement from both male and female patients to follow the risk management program established for the prevention of pregnancy, including double methods for contraception and beta-HCG tests for women of childbearing potential and contraception for males.
* Adequate organ function, including heart, liver, kidney (serum creatinine less than 2 mg/dL)
* Platelet count at least 70 x 10/mcL and absolute neutrophil count at least 1 x 10/mcl

Exclusion criteria:

* Diagnosis of asymptomatic MM or of MGUS based on standard criteria.
* Diagnosis of non-secretory MM.
* Diagnosis of AL Amyloidosis.
* Prior or current systemic therapy for MM, including steroids (with exception of bisphosphonates).
* Patient has received other investigational drugs within 30 days before enrollment.
* Female subjects pregnant or breastfeeding
* Patient has Grade 2 or higher peripheral neuropathy (NCI criteria).
* Patient has a prior history of thrombosis or venous thromboembolism or pulmonary embolism.
* Patient has a previous diagnosis of antiphospholipid antibodies or lupus anticoagulant, factor V Leiden mutation, prothrombin G21210A mutation, antithrombin, protein C or S deficiency.
* Patient has a clear indication to receive a specific other anti-platelet therapy (e.g. clopidogrel, ticlopidine).
* Patient has a clear indication to receive long-term anticoagulant therapy (e.g. prosthetic heart valve, atrial fibrillation).
* Active bleeding or high risk of bleeding (gastrointestinal bleeding within the past 12 months; endoscopic diagnosis of peptic ulcer disease or ulcerative esophagitis within the past 6 months unless there is documented endoscopic evidence of healing; intracranial bleeding within the past year; amyloidosis; known bleeding diathesis).
* Seropositive for HIV, or active hepatitis A, B or C infection.
* Poorly controlled hypertension or diabetes mellitus (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before the start of therapy) or other serious medical or psychiatric conditions that could interfere with adherence to or completion of this study.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Previous or concurrent malignancies at other sites, with the exception of appropriately treated localized epithelial skin or cervical cancer. Patients with remote histories (>5 years) of other cured tumors may be entered.
* Receipt of extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks before enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of CR+nCR to induction treatment | 63 days after the start day of either TD or VTD as induction therapy
  Responses to induction therapy were reported by study investigators and centrally reassessed by study coordinator(s). Criteria are those initially proposed by the European Group for Blood and Marrow Transplantation (EBMT), with the addition of nCR (100% M-protein reduction by electrophoresis, but immunofixation-positive) and very good partial response (VGPR) (at least 90% serum and urine M-protein reduction) categories. Comparisons of response rates between treatment arms are performed using Fisher's exact test.

SECONDARY OUTCOMES:
Rate of CR+nCR to autotransplantation(s) and subsequent consolidation therapy | 90 days after the second autologous transplantation and 70 days after the beginning of either TD or VTD as consolidation therapy
  Responses to autotransplantation(s) and consolidation therapy were reported by study investigators and centrally reassessed by study coordinator(s). Criteria are those initially proposed by the EBMT, with the addition of nCR and VGPR categories. Comparisons of response rates between treatment arms are performed using Fisher's exact test. Comparisons of response rates between treatment arms are performed using Fisher's exact test.
Time To Progression (TTP) | Average time period between the start day of either TD or VTD as induction therapy and the day of relapse or progression
  TTP is defined as time from start of induction treatment with either TD or VTD to relapse or progression, as evaluated according to EBMT criteria. Comparison of TTP between treatment arms is performed using the log-rank test; distributions are estimated using Kaplan-Meier methodology.
Progression-Free Survival (PFS) | Average time period between the start day of either TD or VTD as induction therapy and the day of relapse or progression or death, whichever occurs firstly
  PFS is defined as time from start of treatment to progression/relapse, or death, whichever occurs firstly. Comparison of PFS between treatment arms is performed using the log-rank test; distributions are estimated using Kaplan-Meier methodology.
Overall Survival (OS) | Average time period between the start day of either TD or VTD as induction therapy and the day of death, due to any cause
  OS is defined as time from start of treatment to death. Comparison of OS between treatment arms is performed using the log-rank test; distributions are estimated using Kaplan-Meier methodology.
Safety | Average time period between the start day of either TD or VTD as induction therapy and the day of any toxicity/adverse event(s) recorded during and after study drug administration
  Safety is monitored until 30 days after the last dose of study drug. Toxicities are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0. Rates of adverse events are compared between treatment arms using the chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Cavo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- AOU di Bologna Policlinico S.Orsola-Malpighi, UO di Ematologia, Bologna, Italy

REFERENCES:
- [Derived] Tacchetti P, Pantani L, Patriarca F, Petrucci MT, Zamagni E, Dozza L, Galli M, Di Raimondo F, Crippa C, Boccadoro M, Barbato S, Tosi P, Narni F, Montefusco V, Testoni N, Spadano A, Terragna C, Pescosta N, Marzocchi G, Cellini C, Galieni P, Ronconi S, Gobbi M, Catalano L, Lazzaro A, De Sabbata G, Cangialosi C, Ciambelli F, Musto P, Elice F, Cavo M; GIMEMA (Gruppo Italiano Malattie Ematologiche dell'Adulto Italian Myeloma Network). Bortezomib, thalidomide, and dexamethasone followed by double autologous haematopoietic stem-cell transplantation for newly diagnosed multiple myeloma (GIMEMA-MMY-3006): long-term follow-up analysis of a randomised phase 3, open-label study. Lancet Haematol. 2020 Dec;7(12):e861-e873. doi: 10.1016/S2352-3026(20)30323-9. PMID 33242443
- [Derived] Zamagni E, Nanni C, Dozza L, Carlier T, Bailly C, Tacchetti P, Versari A, Chauvie S, Gallamini A, Gamberi B, Caillot D, Patriarca F, Macro M, Boccadoro M, Garderet L, Barbato S, Fanti S, Perrot A, Gay F, Sonneveld P, Karlin L, Cavo M, Bodet-Milin C, Moreau P, Kraeber-Bodere F. Standardization of 18F-FDG-PET/CT According to Deauville Criteria for Metabolic Complete Response Definition in Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2021 Jan 10;39(2):116-125. doi: 10.1200/JCO.20.00386. Epub 2020 Nov 5. PMID 33151787
- [Derived] Jamet B, Morvan L, Nanni C, Michaud AV, Bailly C, Chauvie S, Moreau P, Touzeau C, Zamagni E, Bodet-Milin C, Kraeber-Bodere F, Mateus D, Carlier T. Random survival forest to predict transplant-eligible newly diagnosed multiple myeloma outcome including FDG-PET radiomics: a combined analysis of two independent prospective European trials. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1005-1015. doi: 10.1007/s00259-020-05049-6. Epub 2020 Oct 2. PMID 33006656
- [Derived] Pezzi A, Cavo M, Biggeri A, Zamagni E, Nanni O. Inverse probability weighting to estimate causal effect of a singular phase in a multiphase randomized clinical trial for multiple myeloma. BMC Med Res Methodol. 2016 Nov 9;16(1):150. doi: 10.1186/s12874-016-0253-9. PMID 27829371
- [Derived] Sonneveld P, Goldschmidt H, Rosinol L, Blade J, Lahuerta JJ, Cavo M, Tacchetti P, Zamagni E, Attal M, Lokhorst HM, Desai A, Cakana A, Liu K, van de Velde H, Esseltine DL, Moreau P. Bortezomib-based versus nonbortezomib-based induction treatment before autologous stem-cell transplantation in patients with previously untreated multiple myeloma: a meta-analysis of phase III randomized, controlled trials. J Clin Oncol. 2013 Sep 10;31(26):3279-87. doi: 10.1200/JCO.2012.48.4626. Epub 2013 Jul 29. PMID 23897961
- [Derived] Cavo M, Pantani L, Petrucci MT, Patriarca F, Zamagni E, Donnarumma D, Crippa C, Boccadoro M, Perrone G, Falcone A, Nozzoli C, Zambello R, Masini L, Furlan A, Brioli A, Derudas D, Ballanti S, Dessanti ML, De Stefano V, Carella AM, Marcatti M, Nozza A, Ferrara F, Callea V, Califano C, Pezzi A, Baraldi A, Grasso M, Musto P, Palumbo A; GIMEMA (Gruppo Italiano Malattie Ematologiche dell'Adulto) Italian Myeloma Network. Bortezomib-thalidomide-dexamethasone is superior to thalidomide-dexamethasone as consolidation therapy after autologous hematopoietic stem cell transplantation in patients with newly diagnosed multiple myeloma. Blood. 2012 Jul 5;120(1):9-19. doi: 10.1182/blood-2012-02-408898. Epub 2012 Apr 12. PMID 22498745
- [Derived] Cavo M, Tacchetti P, Patriarca F, Petrucci MT, Pantani L, Galli M, Di Raimondo F, Crippa C, Zamagni E, Palumbo A, Offidani M, Corradini P, Narni F, Spadano A, Pescosta N, Deliliers GL, Ledda A, Cellini C, Caravita T, Tosi P, Baccarani M; GIMEMA Italian Myeloma Network. Bortezomib with thalidomide plus dexamethasone compared with thalidomide plus dexamethasone as induction therapy before, and consolidation therapy after, double autologous stem-cell transplantation in newly diagnosed multiple myeloma: a randomised phase 3 study. Lancet. 2010 Dec 18;376(9758):2075-85. doi: 10.1016/S0140-6736(10)61424-9. Epub 2010 Dec 9. PMID 21146205